CLINICAL TRIAL: NCT01481233
Title: Phase II Trial of Oral Colchicine in Men With Castrate-Resistant Prostate Cancer Who Have Failed Taxotere-Based Chemotherapy
Brief Title: Oral Colchicine in Men With Castrate Resistant Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to funding
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Drabick, Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSHCI 09-023
Record Dates: First submitted 2011-11-11; First posted 2011-11-29 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Prostate Cancer
Keywords: oral colchicine; castrate-resistant prostate cancer; failed taxotere based chemotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): Colchicine 0.5 mg BID x 21 days
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — Colchicine 0.6 mg bid to a maximum of 1.2 mg bid
  Other Names: Colcrys

SUMMARY:
The purpose of this study is to determine the prostate specific antigen response to continuous low dose oral colchicine.

DETAILED DESCRIPTION:
The investigators propose a simple phase II trial of oral colchicine at the standard prophylactic dose utilized for gout in men with CRPCa who have failed taxotere based chemotherapy. The investigators will utilize a simple modified Simon 2-stage design. The investigators plan to enroll 40 men for the study. The men should have completed prior taxotere based therapy or any other therapy post-taxotere including cabazitaxel one month prior to receipt of colchicine on trial. Staging with a baseline bone scan, CT and PSA as well as routine CBC, CMP and PAP. The dose of the drug can be escalated as tolerated to a maximum of 1.2 mg bid. The patient would be seen at 21 day intervals. After every 3 cycles of treatment, patient would be restaged with CT and bone scan. Patients with stable disease, partial response or complete response would continue therapy until either disease progression or intolerable toxicity after which the patient would be taken off study.

ELIGIBILITY:
Inclusion Criteria:

* Castrate resistant prostate cancer
* Failure or intolerance of taxotere or cabazitaxel-based chemotherapy or abiraterone administered for castrate resistant prostate cancer is allowed
* Age > 18 years and ability to provide informed consent
* ECOG performance status of 0, 1 or 2
* No prior use of colchicine within the last 2 years
* No chemotherapy, hormonal therapy, immunotherapy or radiation therapy within 1 month of day 1, cycle 1

Exclusion Criteria:

* Inability to provide informed consent
* Hypersensitivity to colchicine
* Severe renal, gastrointestinal or hepatic disorders
* Pre-existing blood dyscrasia
* PLT < 100K, ANC < 1000
* Serum Cr > 2 x ULN
* Bilirubin > 2 ULN
* AST > 2 x ULN
* Concurrent use of CYP3A4 inhibitors which may increase drug levels and toxicity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
PSA Response rate | 63 days (3 cycles of treatment)
  Determine the PSA response rate to continuous low dose oral colchicine

SECONDARY OUTCOMES:
Response rate | 63 days (3 cycles)
  Determine the progression free survival
Toxicity grading | One year
  Determine the safety and tolerability of continuous low dose oral colchicine

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Drabick, MD, Principal Investigator — Milton S. Hershey Medical Center